CLINICAL TRIAL: NCT03580850
Title: INTEREST OF INTRAVENOUS INJECTION OF GADOLINIUM IN EXPLORATION INTRA-LABYRINTHINE SCHWANNOMA IN MRI 3 TESLAS
Brief Title: MRI Scan and Intra-labyrinthine Schwannoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6809
Record Dates: First submitted 2018-02-26; First posted 2018-07-09 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-02

CONDITIONS: Schwannoma
Keywords: intra labyrinthine schwannoma; schwannoma; magnetic resonance imaging (MRI); gadolinium; T2 weighted gradient echo
MeSH Terms: conditions — Neurilemmoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention in this restrospective study — This study is an obervational study

SUMMARY:
Evaluate the interest of gadolinium for the positive and topographic diagnosis of intra-labyrinthine schwannoma, comparing T1 sequence acquired after gadolinium injection to a sequence of fast imaging type employing steady state acquisition (FIESTA-C)

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Have intra-labyrinthine schwannoma
* Have benefited from an MRI with gadolinium injection on the MRI 3T with interpretable sequences of good quality
* Subject giving their consent for their participation
* Subjects who benefited, between 2009 and 2016, from an MRI of the external auditory canals, with gadolinous product injection and on the 3 Tesla MRI, in which a diagnosis of intra labyrinthine schwannoma was made

Exclusion Criteria:

- Refusal to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient having intra-labyrinthine schwannoma
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of intra labyrinthine vestibular nerve tumor using T2 FIESTA alone | 1 hour after the realization of the MRI

CONTACTS AND LOCATIONS:
Overall Officials: Francis VEILLON, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service Imagerie 1, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No